CLINICAL TRIAL: NCT06381557
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Study on the Effectiveness and Safety of Zhengyuan Capsules for Cancer-related Fatigue in Patients With Breast Cancer
Brief Title: Cancer-related Fatigue in Patients With Breast Cancer Treatment With Zhengyuan Capsules
Acronym: CRF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qiang Fu (Other)
Collaborators: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Qiang Fu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: YRPG-PMS-ZYJN-RCT-2022-01
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cancer-related Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: Zhengyuan Capsules
- Control Group (Placebo Comparator)
  Interventions: Drug: Placebo contains 5%-10% Zhengyuan Capsule total mixed powder

INTERVENTIONS:
Drug: Zhengyuan Capsules — Zhengyuan capsules, 4 capsules at a time, 3 times per day;
  Other Names: A listed Chinese Medicine
  Arms: Experimental Group
Drug: Placebo contains 5%-10% Zhengyuan Capsule total mixed powder — Zhengyuan capsules simulator（Placebo contains 5%-10% Zhengyuan Capsule total mixed powder）, 4 capsules at a time, 3 times per day;
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
Traditional Chinese medicine（TCM） has achieved some meaningful results in improving the symptoms and quality of life of cancer patients, but many research results need to be further verified by clinical trials with larger samples and better design.This study aims to investigate effectiveness and safety of Zhengyuan Capsules for cancer-related fatigue in patients with breast cancer.

DETAILED DESCRIPTION:
By conducting multi-center, randomized, double-blind, placebo-controlled clinical research to investigate effectiveness and safety of Zhengyuan Capsules for cancer-related fatigue in patients with breast cancer.This test choose the improvement of fatigue degree as key indicator, and choose the improvement both symptoms of patients and quality of life as second indicators. And last, the study will try to verify its safety and efficacy with some haematological indexs and reveal its mechanism from the perspectives of Cytokines and immunological indicators, so as to explore the advantages of traditional Chinese medicine（TCM） in the treatment of CRF and support some high quality, internationally recognized clinical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or cytologically confirmed as breast cancer; AJCC 8th edition staging for breast cancer is stages I to III, clinically and radiologically confirmed with no tumor recurrence or metastasis.
2. Completed anti-tumor treatment (surgery, radiotherapy, chemotherapy, targeted therapy) for at least 2 months, with no planned anti-tumor treatment during the study period, excluding endocrine therapy.
3. Meets the diagnosis criteria for cancer-related fatigue.
4. Average score on the Brief Fatigue Inventory (BFI) in the 14 days preceding enrollment is ≥4.
5. Life expectancy of at least 6 months.
6. Age between 18 and 70 years old.
7. Patients and their families understand the basic details of the study, agree to cooperate in completing the relevant research; the patient can communicate verbally and in writing; voluntary signing of the informed consent form.

Exclusion Criteria:

1. Presence of significant liver or kidney dysfunction (e.g., alanine transaminase, aspartate transaminase greater than 3 times the upper limit of normal, blood creatinine greater than 1.5 times the upper limit of normal, eGFR &lt;60 mL/min/1.73m²) or abnormalities in the hematological system (platelet count &lt;75×10⁹/L, hemoglobin &lt;100g/L, or neutrophil count &lt;1.5×10⁹/L);
2. Presence of severe primary diseases in the cardiovascular, cerebrovascular, immune systems, or requiring treatment for mental illness;
3. Hypokalemia (blood potassium &lt;3.0mmol/L) or electrolyte imbalance with related symptoms or symptoms that may occur after enrollment;
4. Unimproved hypothyroidism;
5. Hypoalbuminemia (blood albumin &lt;30g/L) or malnutrition (Body Mass Index, BMI &lt;18 kg/m²);
6. Traditional Chinese medicine syndrome pattern consistent with Yin deficiency and internal heat;
7. Use of medications indicated in the instructions or with main functions that meet the following conditions: other Western or Chinese medicine preparations that affect the efficacy evaluation of cancer-related fatigue; undergoing treatment with anti-anemia, anti-anxiety/depression, anti-insomnia, or other psychostimulant drugs; use of drugs with leukocyte-increasing effects within the past week, such as granulocyte colony-stimulating factor (G-CSF);
8. Known allergy to the investigational drug or its components;
9. Breastfeeding, pregnant, or planning to become pregnant within 3 months;
10. The investigator deems the individual unsuitable for participation in this clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue degree with the Brief Fatigue Inventory（BFI） | 8 weeks
  BFI consists of 9 items, each rated from 0 to 10, with fatigue score calculated as the total score divided by 9. A higher score indicates a greater level of fatigue; where 0 indicates no fatigue, 1-3 indicates mild fatigue, 4-6 indicates moderate fatigue, 7-9 indicates severe fatigue, and 10 indicates the most severe fatigue imaginable.In the screening phase, the subjects' fatigue status is assessed using the Brief Fatigue Inventory (BFI). Subjects are required to complete the BFI assessment at a specified time each day for 14 consecutive days and record the assessment results. The Investigators determine the eligibility of subjects based on the average BFI scores over the 14 days, with subjects considered eligible if the BFI average is ≥4 points. During the treatment phase, subjects undergo BFI assessments once a week at specified times (i.e., week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8,) to evaluate their fatigue status.

SECONDARY OUTCOMES:
Fatigue degree the Revised Piper Fatigue Scale（PFS⁃R） | 8 weeks
  PFS-R is derived from the Piper Fatigue Scale by reducing the number of items. It includes 22 items assessing behavior, emotion, sensation, and cognition. Each question is cored from 0 to10 points, where a higher score indicates severe symptoms; 1 to 3 point is mild, 4 to 6 point is moderate, and 7 to 10 point is severe. , resulting in a total fatigue score ranging from 0 to 220. The average score is calculated by dividing the total score by 22. A higher score indicates greater fatigue.Treatment follow-up: Subjects are required to visit the clinic for Visit 3 (4 weeks ± 3 days after medication) and Visit 5 (8 weeks ± 3 days after medication). For Visit 1 (1 week ± 1 day after medication), Visit 2 (2 weeks ± 1 day after medication), and Visit 4 (6 weeks ± 1 day after medication), researchers will conduct follow-up via telephone to assess the subject's condition, encourage, and assist in completing the assessment and recording of the PFS-R scale.
Fatigue degree with the MD Anderson Symptom Inventory（MDASI） | 8 weeks
  MDASI is used to assess various symptoms and discomfort experienced by cancer patients during their treatment. Each question is cored from 0 to10 points, where 0 indicates no symptoms or symptoms without interference, and 10 indicates symptoms reaching the most severe imaginable level and causing severe interference. A higher total score indicates more severe symptoms and higher distress from symptoms.Treatment follow-up: Subjects are required to visit the clinic for Visit 3 (4 weeks ± 3 days after medication) and Visit 5 (8 weeks ± 3 days after medication). For Visit 1 (1 week ± 1 day after medication), Visit 2 (2 weeks ± 1 day after medication), and Visit 4 (6 weeks ± 1 day after medication), researchers will conduct follow-up via telephone to assess the subject's condition, encourage, and assist in completing the assessment and recording of the MDASI scale.
Change of patients' functional status with Karnofsky performance status (KPS) | 8 weeks
  KPS Scores ranged from 100 to 0,The higher score represent the better health, the more likely that you are able to tolerate the side effects of treatment. It is generally considered that Karnofsky80 score or above represent patients can live independently, 60~80 score represent semi-independently, Under 60 represent patients often need help in living.KPS scores should be measured at the baseline, 4 weeks, 8 weeks.
Quality of Life Questionnaire-Breast Cancer Module 23（QLQ-BR23） | 8 weeks
  The EORTC QLQ-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss.Each question is cored from 0 to 4points, where 0 indicates no symptoms or symptoms without interference, and 4 indicates symptoms reaching the most severe imaginable level and causing severe interference. QLQ-BR23 were recorded at the baseline and 8 weeks.

OTHER OUTCOMES:
Adverse reaction rates, including the damage of liver and renal functions that reflected by increased alanine aminotransferase, aspartate aminotransferase and creatinine urea nitrogen respectively | 8 weeks
  Safety evaluation，For Visit 3 (4 weeks ± 3 days after medication), it is mandated to perform the specified examinations. The absence of these tests does constitute a deviation from the protocol. If patients undergo relevant examinations during the course of diagnosis and treatment, the data will be collected.

IPD SHARING:
Plan to Share IPD: No